CLINICAL TRIAL: NCT04322370
Title: Prospective Randomized Blinded Trial of VersaWrap Tendon Protector for Zone 2 Flexor Tendon Injuries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201903272; OCR32662 (Other: University of Florida OnCore)
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Flexor Tendon

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The Occupational hand therapists will be blinded to the use of VersaWrap.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group A (Active Comparator): VersaWrap Treatment Arm- Zone 2 flexor tendon repair with the use of VersaWrap
  Interventions: Procedure: Standard of Care Surgical Procedure; Device: VersaWrap Treatment
- Group B (Active Comparator): Standard of Care Treatment Arm- Zone 2 flexor tendon repair
  Interventions: Procedure: Standard of Care Surgical Procedure

INTERVENTIONS:
Procedure: Standard of Care Surgical Procedure — Zone 2 Flexor Tendon surgical repair will be performed by the principal investigator per standard of care. The same technique of tendon repair will be performed for all patients.
Device: VersaWrap Treatment — is intended to manage and protect tendon injuries where there is no significant loss of tendon tissue
  Arms: Group A

SUMMARY:
To analyze outcomes between patients with Z2FT injuries following repair, randomized to two groups. The first group will be the negative control, with no tendon wrap. The second group will have a VersaWrap Tendon Protector applied over the site of the tendon repair. VersaWrap is current SOC at UF.

DETAILED DESCRIPTION:
VersaWrap Tendon Protector is intended to manage and protect tendon injuries where there is no significant loss of tendon tissue. It functions by separating the healing tendon from surrounding tissues to facilitate tendon gliding and tendon healing. VersaWrap can be placed on, over, or around flexor tendons and remains in place until healing is complete and then is bioresorbed. VersaWrap is FDA cleared for the use in procedures where there is no significant loss of tendon tissue and is currently one of the standard of care treatments used for this injury at UF Health.

VersaWrap Tendon Protector includes a bioresorbable hydrogel sheet and a wetting solution. The sheet is transparent, flexible, ultrathin, non-sided, and can be cut to the desired size. It is made of polysaccharides alginate and hyaluronic acid.

Tendon adhesions are a major problem following repair, particularly for zone 2 flexor tendon (Z2FT) lacerations. The purpose of this study is to prospectively analyze outcomes between patients with Z2FT injuries following repair, randomized to two groups. The first group will be the negative control, with no tendon wrap. The second group will have a VersaWrap Tendon Protector applied over the site of the tendon repair. Outcomes will be evaluated during standard of care post-operative clinic visits at 2 (+/-10 days) weeks, 6 weeks (+/-2 weeks) and 3 months (+/- 1 month) following surgery. Data will be collected from standard of care measurements that include the following outcome measures that will be performed at each follow up visit: range of motion of the affected finger at different joints; total active motion (TAM) of the finger; Strickland modification of TAM (only including proximal interphalangeal (PIP); and distal interphalangeal (DIP) joints), as well as, DASH score and Michigan Hand Outcomes questionnaire. A measurement of grip strength will be obtained at the 3 month follow up visit. This is an important study as adhesions are a particularly serious problem following repair of Z2FT injuries, which can result in persistent finger stiffness and decreased range of motion reducing the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients presenting to the plastic surgery service with a zone 2 flexor tendon injury requiring surgical repair

Exclusion Criteria:

* Patients with a sensitivity or allergy to polysaccharides alginate, hyaluronic acid, or citrate

  * Patients with psychiatric or medical problems that preclude them from having surgery
  * Female patients that are pregnant or breastfeeding
  * Prisoners
  * Patients who are unwilling or unable to follow-up

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-08-21 (Actual); Primary Completion 2027-05-17 (Estimated); Study Completion 2027-05-17 (Estimated)

PRIMARY OUTCOMES:
Strickland modified Total Active Motion (TAM) | At 3 months
  This is an objective assessment of range of motion of the finger (physiological parameter)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Satteson, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No